CLINICAL TRIAL: NCT00005226
Title: Epidemiology of Plasma Fatty Acids and Atherosclerosis
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1106; R01HL040848 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To measure by gas-liquid chromatography the relative concentrations of all saturated and unsaturated fatty acids found in the cholesterol ester and phospholipid fractions of plasma from 4,000 subjects participating in the Atherosclerosis Risk in Communities (ARIC) study. The data were used to clarify the role of various fatty acids in atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

The ARIC study is a large population-based, prospective, multicenter study supported by NHLBI which began in 1986, and is designed to investigate the etiology and natural history of atherosclerosis and cardiovascular risk factors. It involves investigation of four cohorts, each with 4,000 adults ages 45 to 65 from four different communities. The study conducts surveillance for hospitalized myocardial infarction, fatal cardiovascular disease, and stroke in its cohorts and of the community from which they are drawn. Events are classified by a Morbidity and Mortality Classification Committee using standardized criteria.

Data collected on the ARIC cohort at baseline included: a clinical history, a physical examination including blood pressure, height, weight, and anthropometry. A second history and physical examination were performed after three years, and annual telephone interviews were conducted in the intervening years. Laboratory studies at baseline and at three years included: electrocardiogram, pulmonary function tests, ultrasonographic examination of both carotids and one popliteal artery for direct visualization of the atherosclerotic process in peripheral large vessels, and numerous blood studies. Certain hemostatic and lipid tests were performed only in 'cases' with ultrasonographically determined carotid atherosclerosis and matched normal 'controls.'

The ARIC clinical history did collect some dietary history using the Willett Questionnaire, and asked a few questions regarding fish consumption. However, specific questions were brief and only semi-quantitative. Direct measurement of plasma fatty acid content as an ancillary study in the Minnesota cohort of the ARIC study gave far more objective information on specific fatty acid consumption and was invaluable in sorting out the true role that various fatty acids play in the prevention of coronary heart disease. Furthermore, measurement of plasma fatty acids in Minnesota ARIC subjects allowed investigation of the relationships between plasma fatty acids composition and the vast amount of laboratory and clinical outcome data which the ARIC study collected. Because the clinical and other laboratory data for each ARIC participant were already available in the computerized data base, a tremendous amount of valuable information was derived on plasma fatty acid relationships with laboratory findings and clinical outcome in a large, randomly selected United States population.

DESIGN NARRATIVE:

The studies were ancillary to the ARIC study. A cross-sectional study examined the association of plasma fatty acids with plasma lipids, hemostatic parameters, and blood pressure. A nested case-control study examined the association of plasma fatty acids in 75 Minnesota cases with carotid atherosclerosis versus 75 normal matched controls. A third study examined the association of plasma fatty acids with incident clinical cardiovascular events, namely myocardial infarction and stroke.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-07; Study Completion 1992-06

REFERENCES:
- [Background] Ma J, Folsom AR, Lewis L, Eckfeldt JH. Relation of plasma phospholipid and cholesterol ester fatty acid composition to carotid artery intima-media thickness: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Clin Nutr. 1997 Feb;65(2):551-9. doi: 10.1093/ajcn/65.2.551. PMID 9022543
- [Background] Ma J, Folsom AR, Eckfeldt JH, Lewis L, Chambless LE. Short- and long-term repeatability of fatty acid composition of human plasma phospholipids and cholesterol esters. The Atherosclerosis Risk in Communities (ARIC) Study Investigators. Am J Clin Nutr. 1995 Sep;62(3):572-8. doi: 10.1093/ajcn/62.3.572. PMID 7661119
- [Background] Ma J, Folsom AR, Shahar E, Eckfeldt JH. Plasma fatty acid composition as an indicator of habitual dietary fat intake in middle-aged adults. The Atherosclerosis Risk in Communities (ARIC) Study Investigators. Am J Clin Nutr. 1995 Sep;62(3):564-71. doi: 10.1093/ajcn/62.3.564. PMID 7661118
- [Background] Folsom AR, Ma J, Eckfeldt JH, Shahar E, Wu KK. Plasma phospholipid fatty acid composition and factor VII coagulant activity. Atherosclerosis. 1994 Dec;111(2):199-207. doi: 10.1016/0021-9150(94)90094-9. PMID 7718022